CLINICAL TRIAL: NCT04994132
Title: A Randomized Phase 3 Trial of Vinorelbine, Dactinomycin, and Cyclophosphamide (VINO-AC) Plus Maintenance Chemotherapy With Vinorelbine and Oral Cyclophosphamide (VINO-CPO) vs Vincristine, Dactinomycin and Cyclophosphamide (VAC) Plus VINO-CPO Maintenance in Patients With High Risk Rhabdomyosarcoma (HR-RMS)
Brief Title: A Study to Compare Early Use of Vinorelbine and Maintenance Therapy for Patients With High Risk Rhabdomyosarcoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARST2031; NCI-2021-06711 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARST2031 (Other: Children's Oncology Group); ARST2031 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2021-07-09; First posted 2021-08-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-03

CONDITIONS: Alveolar Rhabdomyosarcoma; Botryoid-Type Embryonal Rhabdomyosarcoma; Embryonal Rhabdomyosarcoma; Metastatic Embryonal Rhabdomyosarcoma; Metastatic Rhabdomyosarcoma; Solid Alveolar Rhabdomyosarcoma; Spindle Cell Rhabdomyosarcoma; Spindle Cell/Sclerosing Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma, Alveolar; Rhabdomyosarcoma, Embryonal; Rhabdomyosarcoma | interventions — Specimen Handling; Biopsy; Cyclophosphamide; Dactinomycin; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Vincristine; Vinorelbine; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (VAC, VINO-CPO) (Experimental): Patients receive vincristine sulfate IV on days 1, 8 and 15 of cycles 1-4, 7, 8, 11, and 12, and day 1 of cycles 5, 6, 9, 10, 13, and 14. Patients also receive dactinomycin IV over 1-15 minutes or IVP over 1-5 minutes on day 1 of cycles 1-5, 8-10, and 11-14, and cyclophosphamide IV over 60 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 14 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on weeks 13 and 40.
  MAINTENANCE: Patients receive vinorelbine tartrate IV over 6-10 minutes on days 1, 8, and 15, and cyclophosphamide PO on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Patients in both arms undergo CT, MRI, PET, x-ray imaging, and/or bone scan, as well as blood sample collection throughout the trial. Patients may also undergo bone marrow aspiration and/or biopsy as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Drug: Vincristine Sulfate; Drug: Vinorelbine Tartrate; Procedure: X-Ray Imaging
- Arm B (vinorelbine, VAC, VINO-CPO) (Experimental): Patients receive vinorelbine tartrate IV over 6-10 minutes on days 1 and 8, vincristine sulfate IV on day 15, dactinomycin IV over 1-15 minutes or IVP over 1-5 minutes on day 1 of cycles 1-5 and 8-14, and cyclophosphamide IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 14 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on weeks 13 and 40.
  MAINTENANCE: Patients receive vinorelbine tartrate IV over 6-10 minutes on days 1, 8, and 15, and cyclophosphamide PO on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Patients in both arms undergo CT, MRI, PET, x-ray imaging, and/or bone scan, as well as blood sample collection throughout the trial. Patients may also undergo bone marrow aspiration and/or biopsy as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy; Drug: Vincristine Sulfate; Drug: Vinorelbine Tartrate; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV or PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Biological: Dactinomycin — Given IV
  Other Names: Actinomycin A IV; Actinomycin C1; Actinomycin D; Actinomycin I1; Actinomycin IV; Actinomycin X 1; Actinomycin-[thr-val-pro-sar-meval]; Cosmegen; DACT; Dactinomycine; Lyovac Cosmegen; Meractinomycin
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
Drug: Vinorelbine Tartrate — Given IV
  Other Names: Biovelbin; Eunades; KW 2307; KW-2307; KW2307; Navelbine; Navelbine Ditartrate; NVB; Vinorelbine Ditartrate
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase III trial compares the safety and effect of adding vinorelbine to vincristine, dactinomycin, and cyclophosphamide (VAC) for the treatment of patients with high risk rhabdomyosarcoma (RMS). High risk refers to cancer that is likely to recur (come back) after treatment or spread to other parts of the body. This study will also examine if adding maintenance therapy after VAC therapy, with or without vinorelbine, will help get rid of the cancer and/or lower the chance that the cancer comes back. Vinorelbine and vincristine are in a class of medications called vinca alkaloids. They work by stopping cancer cells from growing and dividing and may kill them. Dactinomycin is a type of antibiotic that is only used in cancer chemotherapy. It works by damaging the cell's deoxyribonucleic acid (DNA) and may kill cancer cells. Cyclophosphamide is in a class of medications called alkylating agents. It works by damaging the cell's DNA and may kill cancer cells. It may also lower the body's immune response. Vinorelbine, vincristine, dactinomycin and cyclophosphamide are chemotherapy medications that work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. This trial may have the potential to eliminate rhabdomyosarcoma for a long time or for the rest of patient's life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare event-free survival (EFS) of patients with high-risk rhabdomyosarcoma (HR-RMS) treated with vinorelbine, dactinomycin and cyclophosphamide (VINO-AC) followed by 24 weeks of vinorelbine and oral cyclophosphamide (VINO-CPO) maintenance therapy to that of patients treated with vincristine, dactinomycin and cyclophosphamide (VAC) followed by 24 weeks of VINO-CPO maintenance therapy.

SECONDARY OBJECTIVES:

I. To assess the safety and feasibility of administering VINO-AC in newly diagnosed patients with HR-RMS.

II. To describe the toxicity experience of patients with HR-RMS treated with VINO-AC compared to VAC.

III. To compare overall survival (OS) of patients with HR-RMS treated with VINO AC followed by 24 weeks of VINO-CPO maintenance therapy to that of patients treated with VAC followed by 24 weeks of VINO-CPO maintenance therapy.

IV. To compare objective radiologic response rates at week 12 between patients with HR-RMS treated with VINO-AC to those treated with VAC.

V. To determine whether the addition of 24 weeks of VINO-CPO maintenance therapy improves EFS in patients with HR-RMS when compared to historical controls.

VI. To determine the association between circulating tumor-derived deoxyribonucleic acid (ctDNA) levels at diagnosis and during initial chemotherapy and event-free survival (EFS) in patients with HR RMS.

VII. To prospectively validate the prognostic impact of genomic variants in HR RMS.

EXPLORATORY OBJECTIVE:

I. To collect serial blood samples and tumor tissue for banking at baseline, during treatment, at the end of therapy, and at the time of progression for future tumor and liquid biopsy studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive vincristine sulfate intravenously (IV) on days 1, 8 and 15 of cycles 1-4, 7, 8, 11, and 12, and day 1 of cycles 5, 6, 9, 10, 13, and 14. Patients also receive dactinomycin IV over 1-15 minutes or IV push (IVP) over 1-5 minutes on day 1 of cycles 1-5, 8-10, and 11-14, and cyclophosphamide IV over 60 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 14 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on weeks 13 and 40.

ARM B: Patients receive vinorelbine tartrate IV over 6-10 minutes on days 1 and 8, vincristine sulfate IV on day 15, dactinomycin IV over 1-15 minutes or IVP over 1-5 minutes on day 1 of cycles 1-5 and 8-14, and cyclophosphamide IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 14 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy on weeks 13 and 40.

MAINTENANCE: All patients receive vinorelbine tartrate IV over 6-10 minutes on days 1, 8, and 15 and cyclophosphamide orally (PO) on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

Patients in both arms undergo computed tomography (CT), magnetic resonance imaging (MRI), positron emission tomography (PET), x-ray imaging, and/or bone scan, as well as blood sample collection throughout the trial. Patients may also undergo bone marrow aspiration and/or biopsy as clinically indicated

After completion of study treatment, patients are followed up every 3 months for year 1, every 4 months for years 2-3, and every 6 months for years 4-5.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be =< 50 years of age at the time of enrollment
* Patients with newly diagnosed RMS of any subtype, except adult-type pleomorphic, based upon institutional histopathologic classification are eligible to enroll on the study based upon stage, group, and age, as below. FOXO1 fusion status must be determined by week 4 (day 28) of therapy. RMS types included under embryonal RMS (ERMS) include those classified in the 1995 International Classification of Rhabdomyosarcoma (ICR) as ERMS (classic, spindle cell, and botryoid variants), which are reclassified in the 2020 World Health Organization (WHO) Classification as ERMS (classic, dense and botryoid variants) and spindle cell/sclerosing RMS (encompassing the historical spindle cell ERMS variant and the newly recognized sclerosing RMS variant). Classification of alveolar RMS (ARMS) in the 2020 WHO Classification is the same as in the ICR and includes classic and solid variants

  * ERMS

    * Stage 4, group IV, >= 10 years of age
  * ARMS

    * Stage 4, group IV Patients will be eligible to remain on protocol therapy based upon stage, group, and age
* Bone marrow metastatic disease is based on morphologic evidence of RMS based on hematoxylin and eosin (H&E) stains. In the absence of morphologic evidence of marrow involvement on H&E, patients with bone marrow involvement detected ONLY by flow cytometry, reverse transcriptase (RT)-polymerase chain reaction (PCR), fluorescence in situ hybridization (FISH), or immunohistochemistry will NOT be considered to have clinical bone marrow involvement for the purposes of this study
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/sex as follows (must be performed within 7 days prior to enrollment):

  * Age; Maximum serum creatinine (mg/dL)
  * 1 month to < 6 months; 0.4 mg/dL (male); 0.4 mg/dL (female)
  * 6 months to < 1 year; 0.5 mg/dL (male); 0.5 mg/dL (female)
  * 1 to < 2 years; 0.6 mg/dL (male); 0.6 mg/dL (female)
  * 2 to < 6 years; 0.8 mg/dL (male); 0.8 mg/dL (female)
  * 6 to < 10 years; 1 mg/dL (male); 1 mg/dL (female)
  * 10 to < 13 years; 1.2 mg/dL (male); 1.2 mg/dL (female)
  * 13 to < 16 years; 1.5 mg/dL (male); 1.4 mg/dL (female)
  * >= 16 years; 1.7 mg/dL (male); 1.4 mg/dL (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (must be performed within 7 days prior to enrollment)

  * If there is evidence of biliary obstruction by tumor, then total bilirubin must be < 3 x ULN for age
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with evidence of uncontrolled infection are not eligible
* RMS that is considered a second malignancy and previous cancer(s) that were treated with chemotherapy and/or radiation. Surgical resection alone of previous cancer(s) is allowed
* Patients with central nervous system involvement of RMS as defined below:

  * Malignant cells detected in cerebrospinal fluid
  * Intra-parenchymal brain metastasis separate and distinct from primary tumor (i.e., direct extension from parameningeal primary tumors is allowed).
  * Diffuse leptomeningeal disease
* Patients who have received any chemotherapy (excluding steroids) and/or radiation therapy for RMS prior to enrollment.

  * Note: the following exception:

    * Patients requiring emergency radiation therapy for RMS. These patients are eligible, provided they are consented to ARST2031 prior to administration of radiation
  * Note: Patients who have received or are receiving chemotherapy or radiation for non-malignant conditions (e.g. autoimmune diseases) are eligible. Patients must discontinue chemotherapy for non-malignant conditions prior to starting protocol therapy
* Vincristine and vinorelbine are sensitive substrates of CYP450 3A4 isozyme. Patients must not have received drugs that are moderate to strong CYP3A4 inhibitors and inducers within 7 days prior to study enrollment
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Time from randomization to an event defined as disease relapse/progression, second malignancy, or death, whichever occurs first, assessed up to 5 years from study enrollment
  Will be estimated using the Kaplan-Meier method and will be compared between the two regimens using a log-rank test.

SECONDARY OUTCOMES:
Overall survival | Time from randomization to death of any cause, assessed up to 5 years from study enrollment
  Will be estimated using the Kaplan-Meier method and will be compared between the therapy groups using a log-rank test.
Radiologic response rate | At week 12 after study enrollment
  Includes both complete response and partial response. Response Evaluation Criteria in Solid Tumors 1.1 criteria will be used to define complete and partial responses. Will be compared between arms using chi square test.
Incidence of adverse events | Up to 5 years from study enrollment
  Adverse events of particular interest including grade 4 hematologic toxicity, grade 2 sinusoidal obstruction syndrome, grade 3 or higher neuropathy and any non-hematologic toxicity that result in delays > 14 days in the delivery of a 21-day cycle of therapy or results in a dose reduction of any chemotherapy drugs.
Feasibility and safety assessed by the adverse events, toxicities and treatment delays | From study enrollment to completion of the initial 12 weeks of therapy
  If more than 40% of patients enrolled in the safety phase experience one or more of the toxicities, the study will be paused, the study team will review the data and determine if an amendment is needed.
  Specifically, toxicities of interest include:
  1. Hematological toxicities that delay the administration of subsequent chemotherapy cycles by more than two weeks.
  2. Grade 2 or higher sinusoidal obstruction syndrome.
  3. Grade 3 or higher neuropathy.
  4. Other Grade 3 or higher non-hematological toxicities that delay the administration of subsequent chemotherapy cycles by more than 2 weeks.
Association between circulating tumor-derived deoxyribonucleic acid (ctDNA) and EFS | Up to 5 years from study enrollment
  Will use Kaplan-Meier methods to calculate EFS, defined as the time from randomization to an event defined as disease relapse/progression, second malignancy, or death, whichever occurs first, for patients with and without detectable ctDNA. Will classify patients as having detectable or undetectable ctDNA at baseline. Will compare EFS between these two groups using a one-sided log-rank test.
Prognostic impact of genomic variants | Up to 5 years from study enrollment
  Will provide descriptive statistics for amplifications in MYCN and mutations in TP53 and MYOD1. Will compare EFS between patients with and without these mutations detected at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Allen-Rhoades, Principal Investigator — Children's Oncology Group
Locations (251):
- United States (229):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Westchester Medical Center, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - Valley Medical Center, Renton, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia